CLINICAL TRIAL: NCT05727592
Title: Effectiveness Of 12-Weeks Brazilian Spinach on Health Outcomes Among Type 2 Diabetes Patients in Hospital Universiti Sains Malaysia
Brief Title: An Intervention Study on the Effect of Brazilian Spinach Supplementation on Health Outcomes Among Type 2 Diabetes Patients in Hospital Universiti Sains Malaysia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Juliana binti Shamsudin, Principal Investigator, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: USM/JEPeM/20120630
Record Dates: First submitted 2022-12-29; First posted 2023-02-14 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Interventional study: parallel, single and non-blinded study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Intervention: Diabetic Brazilian spinach supplementation group Subjects in this group will be receiving Brazilian spinach for 12 weeks in which they must consume 15g of Brazilian spinach daily with lunch or dinner.
  Interventions: Dietary Supplement: Althernanthera Sissoo
- Control Group (Experimental): No intervention: Diabetic control group Subjects in this group will not receive Brazilian spinach. However, they will be receiving standard dietary counselling and educated for the same lifestyle intervention as in the intervention group.
  Interventions: Behavioral: Dietary Consultation

INTERVENTIONS:
Dietary Supplement: Althernanthera Sissoo — 15g of Althernanthera Sissoo consumed with lunch or dinner per day.
  Other Names: Brazilian Spinach
  Arms: Intervention Group
Behavioral: Dietary Consultation — Dietary consultation to improve the intakes of vegetables daily
  Arms: Control Group

SUMMARY:
The purpose of this study is to determine whether Brazilian spinach supplementation effective in improving the nutritional status of Type 2 Diabetes Mellitus patient.

DETAILED DESCRIPTION:
Background: Vegetables are valuable health promotion foods because they contain vital nutrients such as vitamins, minerals, proteins, fibres and bio-functional components but are low in fat, sodium and calories as compared with many other foods. In terms of body fat, increase vegetable intake that consist of dietary fibre can play an important role in the regulation of body weight. Therefore, the supplementation of dietary fibre intake from vegetable may have benefit in reducing the percentages of body fat. Though, the clinical effect in human remains unclear and currently no study conducted in Malaysia regarding the effectiveness of this plant towards blood sugar control. Apart from that, lower intake of vegetable among Malaysian, lower cost vegetable choices and higher availability of Althernanthera Sissoo (Brazilian Spinach) due to easy growth may benefit the diabetes patient. Therefore, the investigators plan to conduct this study to determine the effectiveness of 12-weeks Brazilian Spinach supplementation on health outcomes among patients with type 2 diabetes especially in Kelantan region. The investigators hypothesized that diabetes patients on supplementation of Brazilian Spinach would have significant differ in terms of anthropometry, biochemical, clinical, and dietary intake compared to control group.

Method: A single-center randomized, controlled, and two-arm parallel design clinical trial will be carried out in Malaysia especially in Kelantan region. This study enrols 100 patients from Hospital Universiti Sains Malaysia (HUSM) diagnosed with type 2 diabetes. Diabetic patients who meet eligibility criteria will be randomly allocated to two groups, which are Brazilian Spinach treatment group and control group. Both groups will be compared on the primary and secondary outcomes at baseline, 3, 6, and 12 weeks.

Discussion: The study will provide insights into the potential beneficial effect of Brazilian Spinach in type 2 diabetic patients. In addition, the therapeutic effect of Brazilian Spinach towards type 2 diabetes will reflect as a change of metabolite profile in serum.

ELIGIBILITY:
Inclusion Criteria:

* Age between 30-65 years old
* Have confirmed diagnosed with type 2 diabetes mellitus of equal or more than 6 months
* HbA1c levels equal or more than 7% (within the last 3 months of recruitment)
* On at least one oral hypoglycemic agent
* Agree not to take other herbal or nutritional supplements for the duration of study.

Exclusion Criteria:

* Unable to tolerate to fiber especially vegetables
* Type 1 diabetes mellitus
* Pregnant
* Insulin treatment
* Severe diabetic complications including end-stage renal diseases, liver diseases or gastrointestinal diseases
* On coagulant therapy (warfarin)

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2023-06-17 (Actual); Study Completion 2023-09-05 (Actual)

PRIMARY OUTCOMES:
Glycaemic control (HbA1c level) | 3 months
  The outcome to be measured are the hbA1c level in which it will be measured in percentage.
Fasting blood glucose | 3 months
  The outcome to be measured are the fasting blood glucose (FBS) in which it will be measured in mmol/L.

SECONDARY OUTCOMES:
Anthropometric measurements | 3 months
  The outcome to be measured are the BMI in which the weight and height will be combined to report BMI in kg/m^2.
Blood pressure | 3 months
  Both pressures, systolic and diastolic will be assessed that will be measured in millimeters of mercury (mmHg).
Dietary Intake | 3 months
  The dietary intake will be measured by conducting the 24-hours dietary recall toward the subjects.
Liver profile | 3 months
  The outcome to be measured is the liver function test (LFT) which include alanine transaminase (ALT), aspartate transaminase (AST), and alkaline phosphatase (ALP). This outcome will be measured in units per liter (U/L).
Renal profile | 3 months
  The outcome to be measured is the renal function test (RFT) to get an estimate of the glomerular filtration rate (GFR), serum creatine, and to check for proteinuria (albuminuria).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universiti Sains Malaysia, Kubang Kerian, Kelantan, Malaysia

IPD SHARING:
Plan to Share IPD: No